CLINICAL TRIAL: NCT01211431
Title: Post-cesarean Pain Control Via Continuous Infusion of Ropivacain et Diclogenac Into the Wound Versus Intathecal Morphine: Comparison of the Quality of Analgesia, Side Effects, and the Incidence of Residual Scar Pain
Brief Title: Post-cesarean Pain Control Via Continuous Infusion of Ropivacain et Diclogenac Into the Wound Versus Intathecal Morphine
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No inclusions.
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AOI/2008/GA-01; 2008-004643-11 (EudraCT Number)
Record Dates: First submitted 2010-09-28; First posted 2010-09-29 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Cesarean Section
Keywords: cesarean section; pain; ropivacain; diclofena; morphine
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reference (Active Comparator): Intrathécale morphine is used for post-cesarean pain control
  Interventions: Drug: Reference
- Experimental (Experimental): A solution including both ropivacain and diclofenac continuously delivered to the wound is used for post-cesarean pain control
  Interventions: Drug: Experimental

INTERVENTIONS:
Drug: Reference — Intrathécale morphine is used for post-cesarean pain control
  Arms: Reference
Drug: Experimental — A solution including both ropivacain and diclofenac continuously delivered to the wound is used for post-cesarean pain control
  Arms: Experimental

SUMMARY:
The goal is to compare the quality of post-cesarean analgesia, the side effects and the incidence of residual scar pain obtained with intrathecal morphine (reference treatment) or with a continuous intra-wound solution including both ropivacain and diclofenac (experimental treatment).

ELIGIBILITY:
Inclusion Criteria:

* single, normally progressing pregancy
* term > 36 weeks amenorrhea
* BMI between 20 and 25 kg/m^2 before pregnancy
* height between 55 and 90 kg
* cesarean section by Joel-Cohen or Pfannenstiel techniques
* patient has signed consent
* patient has social security coverage

Exclusion Criteria:

* Multiple pregnancy
* pathological pregnancy: hypertension (>140/90 mmHg found during the pregnancy), pre-eclampsia, gestational diabetes
* term < 36 weeks amenorrhea
* non-pregnancy related maternal pathology (insufficiency)
* obesity (BMI > 25 kg/m^2 before pregnancy)
* height < 155 cm or > 180 cm
* weight < 55 kg or > 90 kg
* patient refuses to sign consent
* surgical technique other than Joel-Cohen or Pfannenstiel
* hepatic insufficiency (prothrombin < 60%)
* contra-indications for rachianesthesia: infection, hemostasis problems (platelets < 80.109/L, prothrombin < 60%, TCA > 40s)
* allergy to local anesthestics
* patient is participating in another study, or has participated in another study within the last 6 months
* patient is under any type of guardianship

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-09; Primary Completion 2012-10 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Primary VAS score | 36 hours post delivery
  The patient is asked to evaluate cesarean-section related pain using a visual analog scale (VAS) score for pain on a scale of 1-10 in a sitting position.

CONTACTS AND LOCATIONS:
Overall Officials: Antoinie Guy Aya, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes